CLINICAL TRIAL: NCT01570465
Title: Prospective Survey on Severe Infections During a Multicenter Study of Risk-adapted, MRD-directed Therapy for Young Adults With Newly Diagnosed Acute Myeloid Leukemia.
Brief Title: Prospective Study on Severe Infections on Acute Myeloid Leukemia (AML) Patients
Acronym: AML1411
Status: Terminated | Type: Observational
Why Stopped: low interest
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: AML1411
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: AML; Adult
Keywords: AML; adult; AML1310 GIMEMA study
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients enrolled in the GIMEMA AML1310 study.: * All patients enrolled in the GIMEMA AML1310 study;
  * Signed written informed consent according to ICH/EU/GCP and national local laws.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Assess the impact of each type of severe infections (SI) over the 24-month overall survival of young patients with newly diagnosed acute myeloid leukemia along a predefined antileukemic treatment strategy.

SUMMARY:
All patients receiving induction, consolidation and salvage chemotherapy, and autologous or allogeneic stem cell transplantation according to a strategy defined in the GIMEMA AML1310 protocol will be prospectively monitored for SI (bacteremia, invasive mycoses, other microbiologically documented bacterial infections, pneumonia, other invasive tissue infections and viral diseases) during each chemotherapy and transplant and the impact of these infections on survival will be evaluated until 24 months from the diagnosis of AML.

DETAILED DESCRIPTION:
Treatment of AML patients during chemotherapy and SCT is frequently complicated by SI which may represent an obstacle to the antileukemic chemotherapy and transplant program. Antimicrobial prophylaxis, diagnostic approaches and antimicrobial therapy should be adapted to the infectious risk of the leukemic population. A crucial problem in the definition of these strategies is represented by the continuous change in the epidemiological patterns of infections as a result of the modification of risk factors in the leukemic population and of the global epidemiology of hospital and community acquired infections. In particular, the emergence of antibiotic resistant pathogens, particularly among gram negative bacteria, represents a serious problem which dramatically impacts on the antibacterial prophylaxis and treatments choices. A continuous epidemiology survey is required in order to better define proper prevention, diagnostic and treatment approaches. A common problem in the infections control in immunocompromised populations is represented by a late epidemiological consciousness. In particular, when new antileukemic strategies are implemented any change in the infectious epidemiology is frequently evidenced later retrospectively, but retrospective studies suffer of several drawbacks in the timely and proper collection of data.

The aim of the AML1310 GIMEMA protocol is to prospectively evaluate in a large population of newly diagnosed young AML patients the effect of a risk-adapted, MDR directed antileukemic strategy which includes chemotherapy and SCT. The objective of the trial is to evaluate the treatment strategy in terms of OS at 24 months and secondary objectives include the response rates and outcome according to clinical and biological characteristics at baseline and along the antileukemic treatment. A further secondary objective of the AML1310 study is the evaluation of the quality of life.

A prospective, longitudinal survey of infectious complications occurring in patients enrolled in the AML1310 study along the entire antileukemic program, as an ancillary observational study, may be a useful tool to evaluate in real-time the epidemiological patterns of infections, their impact on the OS, on the antileukemic treatment schedule, and on the quality of life. First, it may allow to assess whether the various types of SI, in addition to well known clinical and leukemia-related prognostic variables, are actually independent prognostic factors for the long-term outcome of AML patients. Second, the results of this survey may offer precious indications for the timely update of the prophylaxis , diagnosis and treatment strategies of infections in AML patients undergoing a modern antileukemic program. The advances in the treatment of AML resulting from the AML1310 study may be further enriched by the epidemiological consciousness derived by a parallel survey of the infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the GIMEMA AML1310 study;
* Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

* Patients not eligible for the GIMEMA AML1310 study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients receiving induction, consolidation and salvage chemotherapy, and autologous or allogeneic stem cell transplantation according to a strategy defined in the GIMEMA AML1310 protocol will be prospectively monitored for SI (bacteremia, invasive mycoses, other microbiologically documented bacterial infections, pneumonia, other invasive tissue infections and viral diseases) during each chemotherapy and transplant and the impact of these infections on survival will be evaluated until 24 months from the diagnosis of AML.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Prognostic role on overall survival | At four years from study entry.
  At 24 months of each type of Severe Infection (SI).

SECONDARY OUTCOMES:
Rate of incidence of SI. | At four years from study entry
  Rate of incidence of SI during chemotherapy, transplantation procedures, and follow up of patients enrolled in the GIMEMA study AML1310
The impact of SI on the respect of the step by step time treatment. | At four years from study entry.
  To estimate the impact of SI on the respect of the step by step time treatment along the GIMEMA study AML1310. SI will be considered among the causes of delay or discontinuation or change of the leukemia treatment schedule.
Risk factors and prognostic factors of each type of SI. | At 4 years from study entry
  To estimate the risk factors and prognostic factors of each type of SI according to baseline leukemia risk (low, intermediate and high risk) as defined in the AML1310 protocol;
Overall and attributable mortality. | At 4 years from study entry.
  To estimate the overall and attributable mortality at 3 months from the onset of the SI. Attributable mortality was defined as progressive organ failure involving the organ(s) in which SI was diagnosed and the absence of other morbid conditions thought, by the attending physician or pathologist, to have contributed to death;
Rate of the in vitro susceptibility pattern to antimicrobials of bacteria causing SI with particular attention to the emerging resistances in gram negative bacteria (ESBL, KPC MDR); | At 4 years from study entry
  To evaluate the rate of the in vitro susceptibility pattern to antimicrobials of bacteria causing SI with particular attention to the emerging resistances in gram negative bacteria (ESBL, KPC MDR);
Rate of patients receiving each type of antibacterial and antifungal prophylaxis strategies employed during the various antileukemic treatments; | At 4 years from study entry
  To evaluate the rate of patients receiving each type of antibacterial and antifungal prophylaxis strategies employed during the various antileukemic treatments;
Rate of antibacterial and antifungal administered treatments guided either empirically or by clinical and microbiological evidences; | At 4 years from study entry
  To estimate the rate of antibacterial and antifungal administered treatments guided either empirically or by clinical and microbiological evidences;
Impact of SI in the quality of life. | At 4 years from study entry
  To evaluate the impact of SI in the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano VENDITTI, Pr., Principal Investigator — Policlinico Tor Vergata di Roma
Locations (46):
- Italy (46):
  - U.O. di Medicina Interna - ASUR Marche 8 - Ospedale Civile, Civitanova Marche, Ancona
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - UO Ematologia con trapianto- AOU Policlinico Consorziale di Bari, Bari
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - U.O.C. di Onco-Ematologia - Centro di Ricerca e Formazione ad Alta tecnologia nelle Scienze Biomediche, Campobasso
  - U.O.C. di Onco-Ematologia - A.O. S.Anna e S.Sebastiano, Caserta
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia C.T.M.O. Istituti Ospitalieri, Cremona
  - Sezione di Ematologia e Fisiopatologia delle Emostasi - Azienda Ospedaliera - Arcispedale S. Anna, Ferrara
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - Ospedale Niguarda ' Ca Granda', Milan
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - Nocera Inferiore U.O. Medicina Interna Ematologia ed Oncologia P.O. Umberto I, Nocera Inferiore
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga, Orbassano
  - U.O. di Oncoematologia -plesso ospedaliero "A. Tortora" di Pagani, Pagani
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale di Piacenza, Piacenza
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Ematologia - Ospedale San Carlo, Potenza
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - A.O. "Sant'Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Padiglione Cesalpino - I piano - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - Policlinico di Tor Vergata, Roma
  - Roma Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - UOC Medicina Trasfusionale e Cellule Staminali Azienda Ospedaliera San Camillo Forlanini, Rome
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari
  - Azienda U.L.S.S.9 - U.O. di Ematologia, Treviso
  - U.O. di Ematologia - Azienda Ospedaliera - Pia Fondazione di Culto e di Religione Card. G.Panico, Tricase
  - Clinica Ematologica - Policlinico Universitario, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation Website — http://www.gimema.it